CLINICAL TRIAL: NCT03470974
Title: National Defense Medical Center
Brief Title: The Effect of Self-Titration and Predictors for Blood Pressure Control in Patients With Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Fung-Wei Chang, Director, Head of Obstetrics and Gynecology, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2-104-05-148
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group receives self-titration strategy training and lifestyle education.
  Interventions: Behavioral: Self-titration strategy
- Control Group (No Intervention): The control group receives usual care and lifestyle education.

INTERVENTIONS:
Behavioral: Self-titration strategy — The self-titration strategy allows patients or medical professionals to adjust their medicine (additional, maintain, or decrease dose) depending on a bespoke plan. The bespoke plan for hypertensive patients involves setting target blood pressure, self-monitoring blood pressure, recording blood pressure readings and constructing a medication titration schedule. Each medication titration step is conducted based on the average home BP measurement readings.
  Arms: Intervention Group

SUMMARY:
This study aims to investigate the relationship among self-efficacy, anxiety, depressive symptoms, quality of life, lifestyle, heart rate variability and blood pressure control; and to examine the effects of self-titration strategy on self-efficacy, anxiety, depressive symptoms,heart rate variability, sodium excretion, lifestyle modification,quality of life, and blood pressure control in patients with hypertension.

DETAILED DESCRIPTION:
Background: Hypertension is the major cause of mortality for the cardiac, vascular and renal disease. The effective control of elevated blood pressure may reduce the damages of several target organs. World Health Organization points out "Innovation and Empowerment for health". The self-titration strategy may empower patients to self-control their diseases, share decision-making and increase their ability to self-management their situations and improve their home blood pressure.

Methods: This experimental study included 222 hypertensive patients from outpatient services of cardiology departments of a medical center in northern Taiwan. We randomly divided the 72 patients into the experimental group (n=111) and control group (n=111). The experimental group received self-titration strategy training and lifestyle modification education; the control group received usual care and lifestyle modification education.

Data were collected for self-efficacy, anxiety symptoms, depressive symptoms, lifestyle and health-related quality of life using self-report questionnaires. Heart rate variability was measured with CheckMyHeart device (DailyCare BioMedical, Chungli, Taiwan). Patients evaluated their home blood pressure by corrected sphygmomanometer. We used the generalized estimating equation to evaluate the effects of the intervention.

Purpose: Primary outcome to evaluate the effects of self-titration strategy on the improvement of home blood pressure in patients with hypertension. Secondary outcomes to evaluate the effects of self-titration strategy on the improvement of self-efficacy, anxiety, depressive symptoms and lifestyle quality of life in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 20 years old.
2. diagnosed with primary hypertension.
3. no addiction to drugs or alcohol.
4. not using anti-depression therapy.
5. able to read and understand Chinese or Taiwanese.
6. willing to participate in this study.

Exclusion Criteria:

1. stroke.
2. arrhythmia.
3. major psychiatric disorders
4. thyroid disease.
5. had received a heart transplant, a permanent pacemaker or an implantable cardioverter defibrillator, diagnosed with (6) cancer, (7) heart failure, or (8) acute myocardial infarction.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
evaluate the effects of self-titration strategy on the improvement of home blood pressure | up to 3 months
  Patients evaluated their home blood pressure by corrected sphygmomanometer.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wen Kao, Ph.D., Study Director — Tri-Service General Hospital
Locations (1):
- Tri-service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kao CW, Chen TY, Cheng SM, Lin WS, Chang YC. A Web-Based Self-Titration Program to Control Blood Pressure in Patients With Primary Hypertension: Randomized Controlled Trial. J Med Internet Res. 2019 Dec 5;21(12):e15836. doi: 10.2196/15836. PMID 31804186